CLINICAL TRIAL: NCT03154957
Title: Management of Acute Dislocation of Emergency in the University Hospital of Strasbourg Shoulder: Retrospective Evaluation of Practices and Proposal of a Clinical Path
Acronym: LuxationsHTP
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6025
Record Dates: First submitted 2017-05-11; First posted 2017-05-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2017-05

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The analysis of professional practices in the emergency department of the Strasbourg CHRU in the management of acute shoulder dislocations aims at proposing a clinical pathway of synthesis taking into account current practices and data from the literature. Thus, the objectives are twofold: first standardize care in emergency rooms and try to improve the weak points of this care.The Investigators will concentrate thier observation work on the medicinal analgesic methods proposed to these patients in order to minimize the pain induced by the external reduction maneuvers performed, in the majority of cases, in the emergencies. This work will ultimately have a real clinical impact on the management of these traumatized patients

ELIGIBILITY:
Inclusion Criteria:

* Adult patient consulting for acute shoulder dislocation

Exclusion Criteria:

* Patient refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient with acute shoulder dislocation
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of shoulder dislocation | Day of consultation of the emergency department

CONTACTS AND LOCATIONS:
Locations (1):
- Service D'Urgences Medico-Chirurgicales Adultes - Htp, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No